CLINICAL TRIAL: NCT04220645
Title: Opportunistic Treatment of Hepatitis C Virus Infection (OPPORTUNI-C): A Pragmatic Clinical Trial of Immediate Versus Outpatient Treatment Initiation Among Hospitalized Patients
Brief Title: Opportunstic Hepatitis C Virus Treatment
Acronym: Opportuni-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Olav Dalgard, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019/128
Record Dates: First submitted 2019-10-01; First posted 2020-01-07 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Hepatitis C; Substance Use Disorders
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Pragmatic clinical trial. Cluster randomised with stepped wedge design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Hospitalised patients with hep C are referred to the outpatient clinic at the medical department following discharge.
  Interventions: Other: Standard of care
- Opportunistic treatment (Experimental): Hospitalised patients with hep C are opportunistically and immediately treated when hospitalized for acute care in psychiatric, addiction treatment or somatic wards
  Interventions: Other: Opportunstic treatment

INTERVENTIONS:
Other: Opportunstic treatment — opportunistically treating HCV infection immediately when hep C patients are hospitalized for acute care in psychiatric, addiction treatment or somatic wards
  Arms: Opportunistic treatment
Other: Standard of care — Referral at discharge
  Arms: Standard of care

SUMMARY:
The project will assess the effect of opportunistically treating hepatitis C virus (HCV) infection immediately when HCV-infected people who inject drugs are hospitalized for acute care in psychiatric, interdisciplinary specialized drug treatment or somatic wards. We will compare this approach with the current standard of care (SOC), which is referral to the outpatient clinic at the medical department following discharge.

DETAILED DESCRIPTION:
The overall objective is to show that opportunistic and immediate administration of HCV treatment is more efficient compared to referral-based SOC. The specific objectives are: 1) to compare the intervention and SOC groups with regards to treatment completion, treatment uptake and virologic response ; 2) to assess the rate of reinfection after successful HCV treatment; and 3) to assess the frequency of resistant associated substitutions before and after virologic treatment failure.

We will use a stepped wedge design and include patients in 7 clusters

Following randomization of the cluster to the immediate treatment, physicians at the participating wards will be notified in writing that for the next time period patients diagnosed with HCV infection should be treated immediately. In addition, lectures presenting the opportunistic approach will be given and the Department of Microbiology will add a brief text to the result of HCV RNA testing reminding about the opportunistic approach. In the medical and the psychiatric departments, consultants from the departments of infectious diseases or gastroenterology will prescribe immediate treatment. In the departments that provide addiction treatment, local physicians will prescribe treatment. Treatment will be prescribed in accordance with current Norwegian treatment recommendations. The intensity of care after discharge will be individualized at the discretion of the treating physician.

ELIGIBILITY:
Inclusion criteria

* Above 18 years of age
* HCV RNA positive
* Inpatient at participating ward
* Signed informed consent must be obtained and documented according to national and local regulations

Exclusion criteria:

* Pregnancy or breastfeeding.
* In involuntarily health care.
* Ongoing treatment of hepatitis C.
* Current participation in another trial that might affect the current study.
* Any reason why, in the opinion of the investigator, the patient should not participate (e.g. not able to comply with study procedures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Treatment completion | 12 weeks
  Proportion in each arm who have been dispensed the last 28 days package of HCV treatment

SECONDARY OUTCOMES:
Sustained virological response | 24 weeks
  HCV RNA undetetctable 12 weeks after end of treatment
Reinfection | Two years
  A HCV RNA strain not present at baseline is detected during or after treatment
End of treatment response | 12 weeks
  Proportion in each arm who have undetectable HCV RNA at the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- AkershusUH, Lørenskog, Select A State Or Province, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Midgard H, Malme KB, Pihl CM, Berg-Pedersen RM, Tanum L, Klundby I, Haug A, Tveter I, Bjornestad R, Olsen IC, Finbraten AK, Dalgard O. Opportunistic Treatment of Hepatitis C Infection Among Hospitalized People Who Inject Drugs (OPPORTUNI-C): A Stepped Wedge Cluster Randomized Trial. Clin Infect Dis. 2024 Mar 20;78(3):582-590. doi: 10.1093/cid/ciad711. PMID 37992203
- [Derived] Midgard H, Finbraten AK, Malme KB, Berg-Pedersen RM, Tanum L, Olsen IC, Bjornestad R, Dalgard O. Opportunistic treatment of hepatitis C virus infection (OPPORTUNI-C): study protocol for a pragmatic stepped wedge cluster randomized trial of immediate versus outpatient treatment initiation among hospitalized people who inject drugs. Trials. 2020 Jun 15;21(1):524. doi: 10.1186/s13063-020-04434-8. PMID 32539853